CLINICAL TRIAL: NCT05526040
Title: Head and Neck Cancer Immunonutrition Supplementation During Cancer Treatment: A Randomized, Open-label Intervention Study
Brief Title: Immunonutrition Supplementation in Head and Neck Cancer Patients Undergoing Cancer Treatment Study
Acronym: HaNIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HaNIS-1
Record Dates: First submitted 2022-08-30; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Head and Neck Cancer
Keywords: immunonutrition; arginine; omega 3 fatty acid; radiotherapy; cancer treatment; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Standard medical nutrition therapy with Immunonutrition
  Interventions: Dietary Supplement: Immunonutrient-enriched oral nutrition supplementation
- Control (Active Comparator): Standard medical nutrition therapy
  Interventions: Dietary Supplement: Standard medical nutrition therapy

INTERVENTIONS:
Dietary Supplement: Immunonutrient-enriched oral nutrition supplementation — Individualized dietary assessment and counselling with additional high energy, high protein, immunonutrient-enriched oral nutrition supplement; taken 3 servings per day, from 1 week prior to cancer treatment and continued throughout the cancer treatment.
  Oral Impact® is an oral nutrition supplement product enriched with arginine (3.3g/sachet), omega-3 fatty acids (0.8g/sachet) and nucleotides (0.3g/sachet). The immunonutrient-enriched formula is also a complete and balanced formula, and is gluten free. The osmolality of the formula is 620 mOsm/kg water.
  Other Names: Oral Impact®, Nestle
  Arms: Intervention
Dietary Supplement: Standard medical nutrition therapy — Individualized dietary assessment and counselling and standard nutrition supplementation via oral nutrition supplementation or enteral nutrition as necessary.
  Arms: Control

SUMMARY:
This is a prospective, randomized, open-label intervention study to evaluate the effectiveness of immunonutrition supplementation in head and neck cancer (HNC) patients during cancer treatment.

DETAILED DESCRIPTION:
The study population will be adult HNC patients receiving radiotherapy and chemotherapy treatment. The targeted number of subjects is 116 patients (58 subjects in each arm). Participants will be randomly assigned to receive standard medical nutrition therapy (individualized dietary assessment and counselling, and standard nutrition supplementation as necessary) or standard medical nutrition therapy with high energy, high protein, immunonutrient-enriched oral nutrition supplementation. Immunonutrition supplementation will begin 1 week prior to cancer treatment and continued throughout the cancer treatment, and to be taken in 3 servings/day. The study involves interviewing of subjects for dietary and nutrition assessment; measurement of weight, body composition, handgrip strength; and data collection from subjects' medical records.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Adult HNC patients, male or female, above 18 years of age
* Primary HNC diagnosis, stage I to III; including: cancer of the nasopharynx, oropharynx, oral cavity, hypopharynx, or larynx, etc.
* Referred and planned for curative-intent cancer treatment (radiotherapy and chemotherapy)
* Eastern Cooperative Oncology Group (ECOG) performance status < 2

Exclusion Criteria:

* Inability or unwillingness to provide written informed consent or comply with the requirements of the protocol
* Patients with metastatic stage or recurring/relapse of cancer at same site
* Planned for palliative cancer treatment
* Underlying severe hepatic failure or renal dysfunction (eGFR < 30ml/min/1.73m2)
* Underlying severe sepsis, neutropenia, immune-deficiencies or autoimmune diseases
* Consumption of supplements or enriched foods containing immunonutrients (omega- 3, arginine or nucleotides) in the previous month prior to study; including dietary supplements such as: fish oil capsules, arginine tablets/powder, RNA capsules, etc.
* Known allergy or intolerance to components of the immunonutrition supplement (cow's milk, fish or soy)
* Enrolment in other cancer treatment trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Body weight (kilograms) | Baseline, weekly review during cancer treatment, 1month post-completion of cancer treatment
  Changes in body weight during study period
Nutrition status - scored Patient-Generated Subjective Global Assessment (PG-SGA) | Baseline, initiation of cancer treatment, completion of cancer treatment, 1month post-completion of cancer treatment
  Changes in nutrition status during study period (3 categories: A- well nourished, B- moderately or suspected of being malnourished, and C- severely malnourished)
Nutrition status - 3-Minute Nutrition Screening (3-minNS) tool | Baseline, initiation of cancer treatment, completion of cancer treatment, 1month post-completion of cancer treatment
  Changes in nutrition status during study period (score of 3 to 4 indicates risk of moderate malnutrition, and score of 5 to 9 indicates risk of severe malnutrition)

SECONDARY OUTCOMES:
Handgrip strength | Baseline, initiation of cancer treatment, completion of cancer treatment, 1month post-completion of cancer treatment
  Changes in handgrip strength during study period
Functional status - Eastern Cooperative Oncology Group (ECOG) Performance Status Score | Baseline, initiation of cancer treatment, completion of cancer treatment, 1month post-completion of cancer treatment
  Changes in functional status during study period (score of 0 to 4; whereby 0- fully active and able to carry out all activities without any restrictions, and 4- completely disabled, unable to carry on any selfcare and confined to bed or chair)

CONTACTS AND LOCATIONS:
Overall Officials: Hazreen Abdul Majid, Prof. Dr., Principal Investigator — Department of Social and Preventive Medicine, Faculty of Medicine, University of Malaya; Sing Ean Tan, Principal Investigator — Department of Social and Preventive Medicine, Faculty of Medicine, University of Malaya
Locations (2):
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No